CLINICAL TRIAL: NCT01158053
Title: A Prospective, Global, Multicenter, Non-Randomized, Non-Blinded Study in Patients With Intermediate Coronary Lesions to Examine the Correlation Between Fractional Flow Reserve (FFR) and Intravascular Ultrasound With Virtual Histology (VH-IVUS)
Brief Title: Vascular Evaluation for Revascularization: Defining the Indications for Coronary Therapy: A Pilot Study
Acronym: VERDICT
Status: Completed | Type: Observational
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: RFC-001
Record Dates: First submitted 2010-06-22; First posted 2010-07-08 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: FFR and VH-IVUS — * Stable Angina(SA), Unstable Angina(UA),Non ST-segment Elevation Myocardial Infarction(NSTEMI) or ST-segment Elevation Myocardial Infarction(STEMI) >48hrs scheduled for cardiac catheterization ± PCI. All patient level inclusion and no exclusion criteria are met Signed Informed Consent
  * No PCI or successful and uncomplicated PCI of all non study lesions. One or more study lesions identified.
  All lesion level inclusion criteria and no exclusion criteria are met.
  * FFR followed by VH-IVUS of study lesion(s)
  * Any additional PCI based on routine clinical practice and FFR/IVUS data?
  * If Yes: Final IVUS with VH imaging, Clinical follow-up at hospital discharge, 30 days, 6 months, and then yearly for 3 years
  * If No: Clinical follow-up at hospital discharge, 30 days, 6 months, and then yearly for 3 years
Device: IVUS and FFR
  Other Names: Eagle Eye IVUS catheter; Prine Wire

SUMMARY:
The present prospective, multicenter study will therefore be performed with the primary objective of establishing the correlation between fractional flow reserve (FFR) and intravascular ultrasound with virtual histology (VH-IVUS)-derived parameters in angiographically intermediate coronary lesions. The current study will also examine the relative prognostic utility of FFR and VH-IVUS as a tool to defer percutaneous coronary intervention (PCI), by assessing the long-term rate (up to 3 years) of lesion-related clinical events if deferred by FFR vs. VH-IVUS versus not deferred PCI.

ELIGIBILITY:
Patient-specific inclusion criteria:

1. Clinical presentation: stable angina, unstable angina, non-ST segment-elevation myocardial infarction (NSTEMI) (Braunwald classification of unstable angina, see Attachment 2) or recent STEMI (>48 hours before enrollment).
2. Patient is scheduled for coronary catheterization with or without percutaneous coronary intervention.
3. Age ≥18 years.
4. Patient is able to read, understand, and sign the informed consent document.
5. Patient agrees to all protocol related procedures, including follow-up through 3 years.

Lesion-specific inclusion criteria:

1. The patient has at least one intermediate coronary lesion to be assessed by FFR and VH-IVUS, defined as a lesion with a visually-estimated diameter stenosis ≥40% to <80% with a visually-estimated angiographic reference segment diameter of 2.75 mm - 4.0 mm.
2. There may only be one study lesion in the major epicardial coronary artery or its branches. All other stenosis in this epicardial coronary artery or its branches must be <40% by visual angiographic assessment. E.g.., if the lesion is in the Left Anterior Descending(LAD), there may be no other significant lesions (≥40%) in the LAD, septals or diagonal branches. A single lesion may have normal or nearly normal appearing segments within the lesion as long as it is contained within one CASS segment. Moreover, a single lesion may span two or more CASS segments as long as there is no normal or nearly normal appearing segments >5mm in length within the lesion. However, if a diseased lesion extends across two or more CASS segments and has one or more >5 mm lengths of normal or nearly normal appearing segments within the lesion, then it is considered 2 separate lesions, and may not be enrolled.
3. More than 1 intermediate lesion per patient may be enrolled, as long as each lesion meets the entry criteria as a study lesion (e.g. one intermediate lesion in 1, 2 or 3 unique epicardial coronary arteries (LAD vs. LCX vs. RCA), with FFR and VH-IVUS performed in each vessel. Thus, up to 3 lesions may be enrolled per patient (one in each major epicardial coronary artery).
4. PCI of any lesion in the target vessel (the main epicardial coronary artery or any of its branches) may not have been performed in the preceding 1 year (including during the index procedure) and may not be planned within the next 1 year.
5. Patients undergoing PCI of non-study lesions in non-study target vessels during the index procedure may be enrolled if one or more qualifying intermediate lesion is otherwise present in a different epicardial vessel, but PCI of all non-study lesions must be performed first (including staged procedures) and must be successful and uncomplicated before formal enrollment into this study. The PCI cannot occur in the epicardial coronary artery or its branches containing the intermediate lesion.

   * Successful PCI is defined as residual diameter stenosis of <50% in all treated lesions with Thrombolysis in Myocardial Infarction (TIMI) -3 flow in all treated vessels.
   * Uncomplicated PCI is defined as the absence of intra-procedural chest pain or ST-segment changes lasting >10 minutes, sustained vessel closure, slow or no reflow, side branch loss, distal embolization, perforation, residual dissection (>type B), or requirement for cardiopulmonary resuscitation, cardioversion or defibrillation, pacemaker insertion, intubation, intra-aortic balloon insertion or intravenous pressors.

Patient-specific exclusion criteria:

1. Prior CABG at any time.
2. The patient is likely to undergo PCI, CABG or other cardiac surgical procedure within 1 year of the procedure.
3. ST-segment elevation myocardial infarction within 48 hours of the procedure.
4. Cardiogenic shock defined as systolic blood pressure <90 mmHg lasting >30 minutes, not responding to intravenous fluids, and/or requiring intravenous pressors or an intra-aortic balloon pump or other hemodynamic support device.
5. Heart failure as defined by New York Heart Association class III or IV (see Attachment 2).
6. Respiratory failure requiring intubation or supplementary oxygen.
7. Left ventricular ejection fraction <30% as determined by 2D echo, nuclear testing, magnetic resonance imaging (MRI), or left ventriculography.
8. Any moderate or severe cardiac valve disease.
9. Cerebrovascular accident or transient ischemic attack (TIA) within the past 60 days, or any permanent neurologic deficit.
10. Chronic renal insufficiency (serum creatinine > 2.5mg/dl).
11. History of drug abuse or alcohol abuse or any other condition making it unlikely that the patient will comply with all study procedures, including follow-up for 3 years
12. Any condition with expected survival <2 years.
13. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following the index procedure. Female patients of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure.
14. Patients currently participating in another study of an investigational drug or device which has not yet reached its primary endpoint.
15. Oral intake by the patient of any caffeinated beverage within 4 hours of the procedure
16. Use within 12 hours of theophylline, aminophylline or any xanthine derivative.

Lesion-specific exclusion criteria:

1. An unprotected left main coronary stenosis is present (visually assessed %DS ≥40%, whether or not requiring treatment). The study lesion cannot be a left main lesion.
2. The intermediate lesion is in a vessel with thrombus, moderate or severe calcification, angulation, or tortuosity. PCI may be performed in such non target vessels or lesions prior to study enrollment, however, as long as successful and uncomplicated, after which the patient is enrolled in the study.
3. The study lesion is an ostial lesion (within 5 mm of the aorta or the distal left main coronary artery) or is bifurcation lesion requiring planned dual stenting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled to undergo a diagnostic cardiac catheterization
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The concordance between FFR and IVUS minimum lumen area(MLA) as assessed by continuous correlation (regression), categorical cutoff values , and being unadjusted and adjusted for lesion length, %plaque burden(PB) and VH-thin capped Fibro Atheroma(TCFA) | 3 year

SECONDARY OUTCOMES:
The concordance between operator assessed % diameter stenosis(DS), core lab assessed %DS, FFR and MLA in intermediate lesions | 3 year
Operator assessed and core lab assessed angiographic %DS, and VH-IVUS MLA, lesion length, %PB, and plaque types in intermediate lesions, with core lab assessment as the reference | 3 year
FFR and VH-IVUS derived MLA, %PB, lesion length, and plaque type in deferred vs. treated lesions | 3 year
Operator revascularization decisions (deferral vs. PCI/coronary artery bypass graft(CABG)) according to operator assessed angiographic %DS, FFR and VH-IVUS results in intermediate coronary lesions | 3 year
Deferred study lesion clinical event rates up to three years according to %DS, FFR and VH-IVUS, and comparison with treated study lesion clinical event rates up to three years | 3 year
Treated study lesion clinical event rates up to three years and their correlation with index FFR and VH-IVUS pre and post stenting | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, MD, Principal Investigator — Columbia University